CLINICAL TRIAL: NCT04389554
Title: Assessment of D-dimer Levels in Pregnant Women Diagnosed With COVID-19
Brief Title: D-dimer Levels in Pregnant With COVID-19
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Merve Aldikactioglu Talmac, MD, Specialist of Obstetrics and Gynecology, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: MTalmac
Record Dates: First submitted 2020-05-14; First posted 2020-05-15 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: COVID-19; D-dimer
Keywords: pregnancy; COVID-19; D-dimer
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Healthy pregnant women
  Interventions: Other: Blood D-dimer assay
- Study Group: Pregnant women with COVID-19
  Interventions: Other: Blood D-dimer assay

INTERVENTIONS:
Other: Blood D-dimer assay — Blood samples will be taken from the patients and will be examined by the ELISA method.

SUMMARY:
D-dimer measurements act as a global indicator of coagulation and activation of fibrinolytic systems. An optimal cut-off value for D-dimer and its effect on prognosis has not yet been assessed to predict mortality in admission. Therefore, studies comparing D-dimer values of COVID-19 patients and healthy pregnant women are needed. Our study gives us the opportunity to make this comparison.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with COVID-19

Exclusion Criteria:

- Having a chronic disease that raises D-dimer levels

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: Kanuni Sultan Suleyman Training and Research Hospital Obstetrics and Gynecology Clinic Patients
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-05-29 (Actual)

PRIMARY OUTCOMES:
Compare D-dimer values of COVID-19 patients and healthy pregnant women | one day

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Turgut Ozal, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Gutierrez Garcia I, Perez Canadas P, Martinez Uriarte J, Garcia Izquierdo O, Angeles Jodar Perez M, Garcia de Guadiana Romualdo L. D-dimer during pregnancy: establishing trimester-specific reference intervals. Scand J Clin Lab Invest. 2018 Oct;78(6):439-442. doi: 10.1080/00365513.2018.1488177. Epub 2018 Jul 5. PMID 29975107